CLINICAL TRIAL: NCT06617988
Title: Investigate Differences in SIRT3 Expression in Granulosa Cells and the Levels of Follicular Fluid Metabolites Among Poor Ovarian Responders Subgroups, and Their Association with IVF Outcomes.
Brief Title: SIRT3 Expression in Granulosa Cells and the Levels of Follicular Fluid Metabolites Among POR Subgroups
Acronym: POR SIRT3
Status: Not yet recruiting | Type: Observational
Sponsor: Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jing-Yan Song, Doctor, Shandong University of Traditional Chinese Medicine
Other Study IDs: SDUTCMPOSEIDONHQS
Record Dates: First submitted 2024-09-23; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Poor Ovarian Response
Keywords: Poor ovarian response; In vitro fertilization and embryo transfer; Sirtuin-3; mRNA expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — Follicular fluid from each participant will be collected on the day of egg retrieval under ultrasound guidance (the fluid is usually discarded in routine clinical practice). Granulosa cells will be separated by centrifugation. All of these biospecimen will be stored at -80°C in the Specimen Bank of the Reproductive and Genetic Department at the Affiliatied Hospital of Shandong University of Traditional Chinese Medicine for future analysis. qRT-PCR will be used to examine the relative expression of SIRT3 in granulosa cells. Specialised kits will be used to detect metabolite levels within the follicular fluid.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Normal prognosis group (control group): Participants included in this group should have normal ovarian reserve: number of antral follicle count ≥5, level of anti-Mullerian hormone ≥1.2 ng/ml, and number of oocytes retrieved in the present IVF-ET cycles>9. All participants in this group receive the standard operation protocol for In vitro fertilization and embryo transfer.
  Interventions: Other: Not applicable- observational study
- Unexpected poor prognosis group: Participants included in this group should have normal ovarian reserve but a poor ovarian response, defined as: number of antral follicle count ≥5, level of anti-Müllerian hormone ≥1.2ng/ml, and number of oocytes retrieved in the present IVF-ET cycles ≤ 9. All participants in this group will receive the standard operation for in vitro fertilization and embryo transfer.
  Interventions: Other: Not applicable- observational study
- Poor prognosis of advanced maternal age group: Participants included in this group are characterized by advanced age (≥35 years) and meet at least one of the following criteria: 1. Number of oocytes retrieved in the current IVF cycle ≤9; 2. Diminished ovarian reserve: level of anti-Mullerian hormone<1.2 ng/ml or number of antral follicle count <5. All participants in this group receive the standard operation protocol for In vitro fertilization and embryo transfer.
  Interventions: Other: Not applicable- observational study
- Expected poor prognosis group: Participants included in this group should have diminished ovarian reserve: number of antral follicle count<5 and level of anti-Mullerian hormone<1.2 ng/ml. All participants in this group receive the standard operation protocol for In vitro fertilization and embryo transfer.
  Interventions: Other: Not applicable- observational study

INTERVENTIONS:
Other: Not applicable- observational study — Not applicable- observational study

SUMMARY:
The goal of this prospective, observational study is to learn about the pathogenesis and biological target of the subtypes of poor ovarian response (POR) during In vitro fertilization and embryo transfer (IVF-ET). The main question it aims to answer is:

1. Can the relative expression level of SIRT3 differentiate between POR subtypes, and do these differences reflect distinct metabolic characteristics among the subtypes?
2. Investigate whether SIRT3 expression levels correlate with clinical outcomes. This study will enroll patients with various POR subtypes and collect discarded follicular fluid and granulosa cells on the day of egg retrieval. IVF outcome information routinely collected in electronic databases will also be recorded. Notably, this is a purely observational study with no additional interventions. Your participation will not alter your clinical treatment compared to other patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women who are married and aged between 20 to 45 years, diagnosed with infertility;
* 2. Individuals undergoing their first or second cycle of in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI), with a scheduled fresh embryo transfer;
* 3. Participants must fulfill the diagnostic criteria corresponding to one of the following prognostic categories as determined by the clinician: Normal prognosis, unexpected poor prognosis, poor prognosis of advanced maternal age, or expected poor prognosis.

Exclusion Criteria:

* 1. A body mass index (BMI) of ≥ 35 kg/m²;
* 2. Participation in cycles involving pre-implantation genetic testing or diagnosis of embryos;
* 3. Involvement in cycles utilizing frozen gametes;
* 4. Engagement in cycles that employ donor-derived oocytes;
* 5. Participation in in vitro maturation cycles;
* 6.The presence of uterine cavity or endometrial abnormalities, including but not limited to fibroids, endometrial polyps, malformations, adenomyomas, endometritis, endometrial thinning, hydrosalpinx, uterine infections;
* 7.The existence of contraindications to assisted reproductive technology or pregnancy, such as uncontrolled liver or kidney dysfunction, diabetes mellitus (with glycated hemoglobin ≤ 7% and fasting blood glucose &lt; 10 mmol/L), hypertension, thyroid disorders, asymptomatic cardiac conditions, moderate-to-severe anemia, malignancies, a history of thromboembolism or thrombosis, severe mental health disorders, acute infections of the urinary and reproductive systems, sexually transmitted infections, and detrimental lifestyle factors including substance abuse. Additionally, exposure to teratogenic levels of radiation, toxins, or medications (such as prednisone, other hormones, adrenaline, antibiotics, or medications for hypertension, cardiovascular issues, or antiviral treatment) during surgical procedures, as well as any physical conditions rendering pregnancy inadvisable, are also considered disqualifying factors.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study cohort will prospectively enroll women undergoing in vitro fertilization and embryo transfer (IVF-ET) treatment at the Department of Reproduction and Genetics, Affiliated Hospital of Shandong University of Traditional Chinese Medicine, from October 2024 to January 2025. This cohort will be stratified into four study groups based on the following criteria in equal proportions. All participants will receive the standard operation protocol for In vitro fertilization and embryo transfer.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-01-18 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
The relative expression level of SIRT3 mRNA of granulosa cells | Detected within three days after oocyte retrieval
  The real-time quantitative PCR methods were used to test the relative expression level of SIRT3 mRNA of granulosa cells of each participant among groups.

SECONDARY OUTCOMES:
Positive pregnancy rate | 2 weeks after the day of embryo transfer
  Serum β-hCG level ≥ 10mIU/mL, 14 days after embryo transfer. [Detected via ELISA]
Embryo implantation rate | 3 weeks after the day of embryo transfer
  The number of intrauterine gestational sacs observed divided by the number of embryos transferred. [Detected via ultrasound]
Clinical pregnancy rate | 4 weeks after the day of embryo transfer
  An intrauterine gestational sac with fetal heartbeat detected by transvaginal ultrasonography. [Detected via ultrasound]
Number of oocytes retrieved | Within 1 day after the oocyte retrieval
  The total number of oocytes retrieved in the In Vitro Fertilization and Embryo transfer cycle.
Average daily dose of gonadotropin per COS cycle | Through the process of controlled ovarian stimulation, an average of 10 days
  Average daily dose of gonadotropin per COS cycle
Total dosage of gonadotropin per COS cycle | Through the process of controlled ovarian stimulation, an average of 10 days
  Total dosage of gonadotropin per COS cycle

OTHER OUTCOMES:
Levels of follicular fluid metabolites | Detected within three days after oocyte retrieval
  Patients will be randomly selected from each group and the levels of metabolites (including lactate, pyruvate, malondialdehyde, glutathione) in the follicular fluid will be measured using the corresponding kits.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Gao Sun, M.D, Principal Investigator — Affiliated Hospital of Shandong University of Traditional Chinese Medicine
Locations (1):
- Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cozzolino M, Herraiz S, Titus S, Roberts L, Romeu M, Peinado I, Scott RT, Pellicer A, Seli E. Transcriptomic landscape of granulosa cells and peripheral blood mononuclear cells in women with PCOS compared to young poor responders and women with normal response. Hum Reprod. 2022 May 30;37(6):1274-1286. doi: 10.1093/humrep/deac069. PMID 35451009
- [Background] Jiang Z, Shi C, Han H, Wang Y, Liang R, Chen X, Shen H. Mitochondria-related changes and metabolic dysfunction in low prognosis patients under the POSEIDON classification. Hum Reprod. 2021 Oct 18;36(11):2904-2915. doi: 10.1093/humrep/deab203. PMID 34545401
- [Background] Wang T, Cao Y, Zheng Q, Tu J, Zhou W, He J, Zhong J, Chen Y, Wang J, Cai R, Zuo Y, Wei B, Fan Q, Yang J, Wu Y, Yi J, Li D, Liu M, Wang C, Zhou A, Li Y, Wu X, Yang W, Chin YE, Chen G, Cheng J. SENP1-Sirt3 Signaling Controls Mitochondrial Protein Acetylation and Metabolism. Mol Cell. 2019 Aug 22;75(4):823-834.e5. doi: 10.1016/j.molcel.2019.06.008. Epub 2019 Jul 10. PMID 31302001
- [Background] Gershon E, Plaks V, Dekel N. Gap junctions in the ovary: expression, localization and function. Mol Cell Endocrinol. 2008 Jan 30;282(1-2):18-25. doi: 10.1016/j.mce.2007.11.001. Epub 2007 Nov 19. PMID 18162286
- [Background] Imanaka S, Shigetomi H, Kobayashi H. Reprogramming of glucose metabolism of cumulus cells and oocytes and its therapeutic significance. Reprod Sci. 2022 Mar;29(3):653-667. doi: 10.1007/s43032-021-00505-6. Epub 2021 Mar 5. PMID 33675030
- [Background] Richani D, Dunning KR, Thompson JG, Gilchrist RB. Metabolic co-dependence of the oocyte and cumulus cells: essential role in determining oocyte developmental competence. Hum Reprod Update. 2021 Jan 4;27(1):27-47. doi: 10.1093/humupd/dmaa043. PMID 33020823
- [Background] Gilchrist RB, Ritter LJ, Armstrong DT. Oocyte-somatic cell interactions during follicle development in mammals. Anim Reprod Sci. 2004 Jul;82-83:431-46. doi: 10.1016/j.anireprosci.2004.05.017. PMID 15271471
- [Background] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Background] Matzuk MM, Lamb DJ. The biology of infertility: research advances and clinical challenges. Nat Med. 2008 Nov;14(11):1197-213. doi: 10.1038/nm.f.1895. Epub 2008 Nov 6. PMID 18989307